CLINICAL TRIAL: NCT07213284
Title: Site Randomized Trial to Evaluate Behavioral Intervention Via Web-Based Application (MI MOM- Michigan Healthy Moms Application) to Improve Pregnancy Outcomes
Brief Title: Michigan Healthy Mom (MI-MOM) Pregnancy Improvement Web Application Trial
Acronym: MI-MOM App
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Professor- Tenure System, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00011005; U54HD113291 (NIH)
Record Dates: First submitted 2025-08-14; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; Pregnancy, Complications; Pregnancy Outcomes
Keywords: Pregnancy; App; Behavioral Intervention; Web-based Application; Postpartum
MeSH Terms: conditions — Pregnancy Complications; Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Primary outcomes will be vital record and Medicaid claims data collected independent of this trial, and direct self-report via online survey software.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI MOM (Experimental): Participants receive app content and text messages with information designed to improve pregnancy outcomes.
  Interventions: Behavioral: MI MOM App
- Treatment as Usual (No Intervention): Data collection for study outcomes only

INTERVENTIONS:
Behavioral: MI MOM App — Participants enrolled in the Michigan Healthy Moms (MI MOM) app will receive initial interactive app content followed by regular text messages with information related to pregnancy health, designed to increase patient awareness of warning signs, help them with self-advocacy, and otherwise improve health in pregnancy and postpartum. They will also have online live chat (text) access to a community healthcare worker who can assist them in enrolling in services to improve their health. They will also have the option of enrolling support persons (partners, family members, close friends, etc.) in the MI MOM app to receive similar information designed to help them support the pregnant participant. Providers at intervention sites will also receive information designed to improve their awareness of techniques for preventing maternal morbidity and mortality.
  Arms: MI MOM

SUMMARY:
The purpose of this research study is to see if using the MI MOM App improves pregnancy and postpartum health. There are two study groups, where one group is "treatment as usual" and the other is the "MI MOM App" group. Both groups will be asked to answer questions about their pregnancy health. Researchers will also retrieve vital records and Medicaid claims information related to pregnancy for both groups. Those in the "MI MOM App" group will receive mobile web app content and text messages with informational links and links to videos and micro-interventions. They will also identify up to three close friends or family members who will be invited to receive text messages. Those in the "MI MOM App" will also have the option to contact a community health worker as needed.

DETAILED DESCRIPTION:
The researchers aim to use a site-randomized design to determine whether the Michigan Healthy Mom (MI MOM) app will improve pregnancy health when used by pregnant women, their supporters (partners, mothers, friends, etc.), and healthcare providers, vs treatment as usual. Specifically, the researchers will test:

1. Whether use of the MI MOM app results in improvements to self-reported app targets (e.g., reducing provider bias, increasing treatment-seeking, service connection, early warning sign awareness, and improving mental health)
2. Whether use of the MI MOM app improved overall pregnancy and postpartum health
3. Whether the app reduced disparities in pregnancy/postpartum health, i.e. between Black and White, rural and urban participants

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at 20 weeks gestation or less
* 18 years of age or older
* Access to smartphone with text messaging and internet access
* Speaks English
* Enrolled in Medicaid for health insurance

Exclusion Criteria:

* Younger than 18 years old
* Not pregnant or pregnant with more than 20 weeks gestation
* No access to a smartphone with text messaging and internet access
* Not English speaking
* Not enrolled in Medicaid for health insurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Total pregnancy-associated morbidity through one year postpartum | Start of pregnancy through 1 year postpartum
  Total pregnancy-associated non-severe and severe maternal morbidity through 1 year postpartum. Non-severe maternal morbidity will be indexed using ICD codes taken from Medicaid records, with conditions taken from World Health Organization-identified Maternal Morbidity conditions (e.g., anemia, hypertension, depression). Severe maternal morbidity will use ICD codes identified for the 21 severe maternal morbidity indicators developed by the CDC.
Pregnancy-Associated Mortality through one year postpartum | Start of Pregnancy through 1 year postpartum
  Total pregnancy-associated mortality through 1 year postpartum as measured using a preexisting linked dataset of Medicaid claims, deaths, birth records, and Evidence-Based Practice Center (EPC) program data.
Composite Index, total number of maternal morbidity and mortality risk factors | Measured at 6 weeks post-baseline, 35 weeks of pregnancy, 6 weeks postpartum, 6 months postpartum, and 1 year postpartum.
  A composite index evaluating multiple maternal morbidity and mortality behavioral risk factors including the Tobacco, Alcohol, Prescription medication, and other Substance use Tool for substance use (TAPS); the Humiliation, Afraid, Rape, Kick questionnaire for intimate partner violence (HARK); the Patient Health Questionnaire (PHQ-9) and Generalized Anxiety Disorder Screener (GAD-7) for symptoms of depression and anxiety; patient understanding of early warning signs of pregnancy complications and appropriate responses; confidence in ability to communicate effectively with healthcare providers; help-seeking behaviors/service utilization, and prenatal care adherence. Total score on this composite index will be the number of risks on which the participant is positive at that assessment point. All risks will refer to the time since becoming pregnant (baseline) or since the last assessment point (follow-up observations) except for depression and anxiety, which refer to the past two weeks.

IPD SHARING:
Plan to Share IPD: Yes
All study data that does not reveal participant identity.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Following NICHD data and specimen hub standards.
Access Criteria: Following NICHD data and specimen hub standards.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Derived] Kelpin SS, Margerison CE, McKay AS, Vickers E, Crawford MK, Spencer J, Sikorskii A, Ondersma SJ. Site-randomised trial of a multilevel digital intervention to reduce maternal morbidity and mortality: a study protocol. BMJ Open. 2025 Dec 21;15(12):e113340. doi: 10.1136/bmjopen-2025-113340. PMID 41423300
- [Derived] Kelpin SS, Margerison CE, McKay AS, Vickers E, Crawford MK, Spencer J, Sikorskii A, Ondersma SJ. A study protocol for a site-randomized trial of a multi-level digital intervention to reduce maternal morbidity & mortality. medRxiv [Preprint]. 2025 Oct 31:2025.10.29.25339066. doi: 10.1101/2025.10.29.25339066. PMID 41282939
- See also: Related Info — https://www.pc-pramm.org/